CLINICAL TRIAL: NCT01597037
Title: Aphasia Rehabilitation: Modulating Cues, Feedback & Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Leora Cherney, Senior Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DC011754 (NIH)
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Speech Rehabilitation
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High complexity, high feedback (Active Comparator): Scripts are one grade level higher than the typical script that would be provided for the severity of aphasia; there is an opportunity for the participant to listen to his/her production and assess performance.
  Interventions: Behavioral: Script training
- High complexity, low feedback (Active Comparator): Scripts are one grade level higher than the typical script that would be provided for the severity of aphasia; there is no opportunity for the participant to listen to his/her production and assess performance.
  Interventions: Behavioral: Script training
- Low complexity, high feedback (Active Comparator): Scripts are one grade level lower than the typical script that would be provided for the severity of aphasia; there is an opportunity for the participant to listen to his/her production and assess performance.
  Interventions: Behavioral: Script training
- Low complexity, low feedback (Active Comparator): Scripts are one grade level lower than the typical script that would be provided for the severity of aphasia; there is no opportunity for the participant to listen to his/her production and assess performance.
  Interventions: Behavioral: Script training

INTERVENTIONS:
Behavioral: Script training — 90 minutes/day, 6 days a week; includes 3 weeks of training

SUMMARY:
The purpose of this study is to evaluate how changing different conditions of the speech-language treatment (such as cues, feedback, complexity and practice schedule) affects the language outcome of study subjects with aphasia (i.e., difficulty with the comprehension and expression of spoken and written language) following a stroke.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the most common cause of disability in the United States. According to the American Stroke Association, the prevalence of stroke in the U.S. is approximately 4.8 million with approximately 700,000 additional strokes occurring annually. Approximately 150,000 to 250,000 stroke survivors becoming severely and permanently disabled each year.

A common neurological deficit among stroke survivors, and thus a substantial contributor to post-stroke disability, is aphasia. The loss of, or difficulty with language is extremely debilitating. Recently, there has been an emphasis on the need for intensive aphasia treatment in order to make the long-term neuroplastic changes associated with recovery. However, specific information regarding effective learning parameters is limited.

A number of variables and practice conditions, deriving from motor learning theory, potentially impact the rehabilitation process. Several of these variables have begun to be addressed in the literature, but with conflicting or scant evidence to date. Variables include the type and degree of external cueing, low versus high feedback conditions, task complexity, and practice distribution and schedule.

The purpose of this study is to:

* Modulate variables of cuing, feedback and script complexity that potentially affect treatment outcomes, and measure their effects on acquisition, maintenance and generalization of script learning. These investigations are conducted as separate studies, with the first study being a cross-over study investigating cuing and the second study being a 2x2 factorial design investigating feedback and complexity.
* Modify and optimize AphasiaScripts-an existing treatment program having experimental support for its efficacy-by incorporating these findings.
* Conduct a clinical trial, incorporating the optimized AphasiaScripts program, in order to measure the effect of massed vs distributed practice, and blocked vs random practice schedules, on the acquisition, maintenance and generalization of script learning.

Measures will include independent pre-and post assessments of acquisition, maintenance and generalization of script learning as well as dependent item/cue level measures of progress.

Results and computational models of acquisition, maintenance and generalization will contribute new evidence to support not just the efficacy and delivery of AphasiaScripts, but also the application of practice principles to aphasia treatment in general.

The first part of the study - a cross-over study that evaluates error-free versus error-reducing script training has been done. Below is a description of the second part of the study which evaluates feedback and script complexity.

ELIGIBILITY:
Inclusion Criteria:

* A single unilateral left-hemisphere stroke
* Aphasia Quotient between 40 and 80 on the Western Aphasia Battery
* Age 21 or older
* At least 6 months post-stroke
* Able to comply with the study protocol
* Premorbidly right-handed, as determined by the Edinburgh Handedness Inventory
* Fluent in English premorbidly
* Completed at least 8th grade education

Exclusion Criteria:

* More than one stroke
* Any other neurological condition that could potentially affect cognition, speech or language.
* Global aphasia or inability to participate in routine speech therapy
* Major active psychiatric illness that may interfere with required study procedures
* Untreated or inadequately treated depression
* Current abuse of alcohol or drugs
* Unable to understand, cooperate or comply with study procedures
* Significant visual or auditory impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2017-09 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Percent accurate script related words | Change from baseline to post-treatment in three weeks
  For trained script, untrained script, generalization script

SECONDARY OUTCOMES:
Rate of script-related words | Change from baseline to post-treatment in three weeks
  For trained script, untrained script, generalization script

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Aphasia Research & Treatment, Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Cherney LR, Van Vuuren S. Complexity and Feedback During Script Training in Aphasia: A Feasibility Study. Arch Phys Med Rehabil. 2022 Jul;103(7S):S205-S214. doi: 10.1016/j.apmr.2022.03.002. Epub 2022 Mar 15. PMID 35304120